CLINICAL TRIAL: NCT02387242
Title: Evaluating Pharmacokinetics and Whole Blood Bactericidal Activity Against Mycobacterium Tuberculosis of Single 'High' Doses of Rifampicin in Healthy Volunteers
Brief Title: Whole Blood Bactericidal Activity (WBA) Against Mycobacterium Tuberculosis of Rifampicin in Healthy Volunteers
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: New relevant data published
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: High Rif-WBA
Record Dates: First submitted 2015-02-24; First posted 2015-03-12 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Whole blood Bactericidal Activity; WBA; Rifampicin
MeSH Terms: conditions — Tuberculosis | interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): 10mg/kg Rifampicin
  Interventions: Drug: Rifampicin
- Group 2 (Experimental): 20mg/kg Rifampicin
  Interventions: Drug: Rifampicin
- Group 3 (Experimental): 30mg/kg Rifampicin
  Interventions: Drug: Rifampicin

INTERVENTIONS:
Drug: Rifampicin — Single oral dose of rifampicin
  Other Names: Rifampin

SUMMARY:
The purpose of this study is to evaluate the bactericidal activity against Mycobacterium tuberculosis of standard and high doses of rifampicin. Pharmacokinetics (PK) and Whole blood Bactericidal Activity (WBA) will be measured in healthy volunteers following a single dose of rifampicin at standard dose (10mg/kg) or at high dose (20mg/kg or 30mg/kg).

DETAILED DESCRIPTION:
WBA is an ex vivo model for measuring the combined effects of administered drugs, host factors and strain factors on mycobacterial killing. If performed in parallel with PK measurements, the method can be used to evaluate the effect of drugs throughout the dosing cycle. This study aims to compare different doses of rifampicin in the WBA model, compare activity of rifampicin on WBA by different mycobacterium tuberculosis strain types and assess the host immune response following drug administration.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 21 and above
2. Male or female willing to comply with the study visits and procedures
3. Willing and able to provide written informed consent

Exclusion Criteria:

1. Women who are currently pregnant or breastfeeding
2. Signs of active TB
3. On immunosuppressant, antibiotic or any medication known to have interaction with rifampicin
4. Previous allergy to Rifampicin
5. Evidence of renal or hepatic dysfunction or any clinically significant deviation from normal during screening including laboratory determinations
6. Known hepatic disease or alcohol abuse
7. Current use of any other drugs, over the counter medications and herbal preparations that are known or potential inhibitors or inducers of cytochrome P450 enzymes
8. Any other significant condition that would, in the opinion of the investigator, compromise the volunteer's safety or outcome in the trial
9. Current participation in other clinical intervention trial or research protocol

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative WBA (reported as change in Mtb log CFU per day) | 24 hours

SECONDARY OUTCOMES:
The pharmacokinetic profile of rifampicin | 24 hours

OTHER OUTCOMES:
Change in host cytokine response after study drug administration | 6 hours following administration
  Impact of host immune response before and after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Paton, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore